CLINICAL TRIAL: NCT02718794
Title: Crossover Study in Simulation-based and Problem-based Learning in Practice Guideline for Difficult Airway Management
Brief Title: Simulation-based and Problem-based Learning for Difficult Airway Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mrs.Parichad Apidechakul, Faculty of Medicine Siriraj Hospital, Siriraj Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 233/2558(EC4)
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Education
Keywords: Simulation Training [I02.903.847]; Problem-Based Learning [F02.463.425.720]; Airway Management [E02.041]

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simulation training first (Experimental): A highly customized interactive medium or program that allows individuals to learn and practice real world activities in an accurate, realistic, safe and secure environment.
  Interventions: Procedure: Simulation training; Procedure: Problem-based learning
- Problem-based learning first (Experimental): Instructional use of examples or cases to teach using problem-solving skills and critical thinking.
  Interventions: Procedure: Simulation training; Procedure: Problem-based learning

INTERVENTIONS:
Procedure: Simulation training — spend 3 hours for each of 10 nurse anesthetist students with 4 scenarios
Procedure: Problem-based learning — spend 3 hours for PBL steps with each of 10 nurse anesthetist students

SUMMARY:
Teaching and learning of difficult airway management are considered to be an essential skill in anesthesiology. As a result, doctors and nurses in anesthesia have to be vigilant in every step including airway assessment, equipment preparation and strategic planning of the process.

During the one-year training program, nurse anesthetist students intensively study theories and practical skills in anesthesia, using manikins to living patients. Difficult airway management has become a distinguished means in the training curriculum. In addition, the educational tool in the anesthesia curriculum is typically simulation-based learning (SBL) and problem-based learning (PBL) courses. As a result, we designed a cross-over study to determine the learning achievement of nurse anesthetist students in difficult airway management. The objectives were to study the learning achievement and relative growth of knowledge of the two learning techniques: SBL and PBL.

Thirty-six nurse anesthetist students in Academic Year 2015, volunteered to join the study project. After signing the consent form, they were randomly put into two groups: A (n = 17) and B (n = 19). As designed by the cross-over study, students in group A attended SBL and after 6 weeks, they focused on PBL, and vice versa for group B.

The 40-item, multiple choices exam was developed in regard to difficult airway management guidelines. The correctness and appropriateness of the test (content validity) were determined by three board-certified anesthesiologists. The try out of the test was performed by 10 novice nurse anesthetists. The index of item objective congruence was 0.82 with Kuder Richardson 21 of 0.8. The assessed criterion-referenced item difficulty and discrimination index were 0.4-0.6 and 0.6-0.8 respectively.

The pretest (X1, X2) were post-test ((Y1, Y2) were performed in the consequence. The relative growth of knowledge (G1, G2) was calculated as follows:

G1 = 100 (Y1 - X1) / (F - X1) % G2 = 100 (Y2 - X2) / (F - X2) %

Where F was the full scores of the learning course

Statistics analysis The test scores and relative growth of knowledge between the two groups were expressed as mean and standard deviation. Comparison between the two groups was performed by repeated measure ANOVA. Statistically significant differences were considered when there was a p value of < 0.05 with a 95% confidence interval.

DETAILED DESCRIPTION:
Introduction Teaching and learning of difficult airway management are considered to be an essential skill in anesthesiology. Assessment of the training program requires a currently established guideline. Recent studies revealed that the management of the airway was the most sophisticated maneuver for all anesthesia providers, since it is related to morbidity and mortality circumstances. It appeared in 6.2% of endotracheal intubations in the operating theater. In addition, difficult intubation with ventilation occurred in 1.5%, of the procedures; impossible intubation and difficult ventilation 0.3 %; and "can't intubate, can't ventilate" (CICV) situation, 0.07%.

Normally, most anesthesia personnel perform endotracheal intubation under general anesthesia. However, they occasionally come across difficult airways. This becomes a life- and-death condition that may lead to uneventful sequelae. In practice, a difficult airway is defined as either troublesome facemask ventilation or tracheal intubation. As a result, doctors and nurses in anesthesia have to be vigilant in every step including airway assessment, equipment preparation and strategic planning of the process. In addition, updated difficult airway algorithm helps them manage the patient's airway at the right time.

After graduation, registered nurses need to spend one more year on a training program to become nurse anesthetists, serving as either an anesthesiologist's assistant or a general practitioner's helper. During the one-year training program, nurse anesthetist students intensively study theories and practical skills in anesthesia, using manikins to living patients. However, effective training in airway management results from the learners' competences and from a diversity of teaching techniques.

Currently, the educational tool in the anesthesia curriculum is typically simulation-based learning (SBL) and problem-based learning (PBL) courses, both of which have been widely accepted in many educational institutes. They yield a promising outcome amongst students of professionalism. The SBL provides high-level learning circumstances to help students gain their experiences. The diagnostic and feedback system help learners correct their mistakes with confidence. However, PBL allows students to present their informative knowledge, resulting in retention and integration of learning with clinical experience. In addition, self-directed learning gives them creative thinking. Instructors act as facilitators who empower students to implement their own strategic plan of learning.

Either SBL or PBL has its unique process to assess participants' core knowledge. Furthermore, difficult airway management has become a distinguished means in the training curriculum. As a result, we designed a cross-over study to determine the learning achievement of nurse anesthetist students in difficult airway management.

Objectives To study the learning achievement and relative growth of knowledge of the two learning techniques: SBL and PBL.

Methods Thirty-six nurse anesthetist students in Academic Year 2015, Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University, volunteered to join the study project without any honorarium. The benefit of taking part in the study was only knowledge and clinical experience gained. The students were informed about the significance of the research under the faculty policy as well as the learning objectives in details. After signing the consent form, they were randomly put into two groups: A (n = 17) and B (n = 19). As designed by the cross-over study, students in group A attended SBL and after 6 weeks, they focused on PBL, and vice versa for group B.

The PBL learning session comprised four different clinical questions together with educational resources for one hour self-study. Consequently, all students spent two more hours on presentation and discussion of knowledge information in front of the class. The SBL learning session consisted of the same clinical scenarios as PBL. All learners spent three hours in the environment of a well-equipped operating theater with a standardized patient or a high-fidelity manikin. Then they joined the debriefing forum given by an attending staff.

The 40-item, multiple choices exam was developed under the table of specifications and knowledge map in regard to difficult airway management guidelines. The paper-pencil test comprised of evaluation of the airway, basic preparation of difficult airway management, strategy of endotracheal intubation and extubation, and follow up care.

The correctness and appropriateness of the test (content validity) were determined by three board-certified anesthesiologists who had at least 10 years of experience in anesthesia and were not involved in the project. The try out of the test was performed by 10 novice nurse anesthetists. The index of item objective congruence was 0.82 with Kuder Richardson 21 of 0.8. The assessed criterion-referenced item difficulty and discrimination index were 0.4-0.6 and 0.6-0.8 respectively.

The pretest (X1, X2) were post-test ((Y1, Y2) were performed in the consequence. The relative growth of knowledge (G1, G2) was calculated as follows:

G1 = 100 (Y1 - X1) / (F - X1) % G2 = 100 (Y2 - X2) / (F - X2) %

Where F was the full scores of the learning course

Statistics analysis The test scores and relative growth of knowledge between the two groups were expressed as mean and standard deviation. Comparison between the two groups was performed by repeated measure ANOVA using the Statistical Package for Social Sciences for Windows, release 18. Statistically significant differences were considered when there was a p value of < 0.05 with a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Nurse anesthetist students in the academic year of 2015

Exclusion Criteria:

* The unwilling nurse anesthetist students in the academic year of 2015

Ages: 24 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Learning achievement | 3 months
  student achievement scores from pretest 1( X1), post-test 1 (Y1) and pretest 2 (X2) , post-test2 (Y2)

OTHER OUTCOMES:
Relative growth of knowledge | 3 months
  The difference between the scores : The relative growth of knowledge (G1, G2) was calculated as follows
  G1 = 100 (Y1 - X1) / (F - X1) % G2 = 100 (Y2 - X2) / (F - X2) % Where F was the full scores of the learning course

CONTACTS AND LOCATIONS:
Overall Officials: Parichad Apidechakul, B.Ns, M.P.A., Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Siriraj hospital
Locations (1):
- Parichad Apidechakul, Nonthaburi, Changwat Nonthaburi, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Result] Lorello GR, Cook DA, Johnson RL, Brydges R. Simulation-based training in anaesthesiology: a systematic review and meta-analysis. Br J Anaesth. 2014 Feb;112(2):231-45. doi: 10.1093/bja/aet414. Epub 2013 Dec 23. PMID 24368556
- [Result] Hesselfeldt R, Kristensen MS, Rasmussen LS. Evaluation of the airway of the SimMan full-scale patient simulator. Acta Anaesthesiol Scand. 2005 Oct;49(9):1339-45. doi: 10.1111/j.1399-6576.2005.00856.x. PMID 16146473
- [Result] Smithburger PL, Kane-Gill SL, Ruby CM, Seybert AL. Comparing effectiveness of 3 learning strategies: simulation-based learning, problem-based learning, and standardized patients. Simul Healthc. 2012 Jun;7(3):141-6. doi: 10.1097/SIH.0b013e31823ee24d. PMID 22293664
- [Result] Steadman RH, Coates WC, Huang YM, Matevosian R, Larmon BR, McCullough L, Ariel D. Simulation-based training is superior to problem-based learning for the acquisition of critical assessment and management skills. Crit Care Med. 2006 Jan;34(1):151-7. doi: 10.1097/01.ccm.0000190619.42013.94. PMID 16374169
- [Result] Komasawa N, Sanuki T, Fujiwara S, Haba M, Ueki R, Kaminoh Y, Minami T. Significance of debriefing methods in simulation-based sedation training courses for medical safety improvement in Japan. Springerplus. 2014 Oct 28;3:637. doi: 10.1186/2193-1801-3-637. eCollection 2014. PMID 25392805
- [Result] Tanaka PP, Pessoa R, Fernandes R, Brodsky J. [What is missing for difficult airway management in the 21st century]. Rev Bras Anestesiol. 2015 May-Jun;65(3):235-6. doi: 10.1016/j.bjan.2013.11.008. Epub 2014 Sep 26. No abstract available. Portuguese. PMID 25990498
- [Result] Ross AJ, Kodate N, Anderson JE, Thomas L, Jaye P. Review of simulation studies in anaesthesia journals, 2001-2010: mapping and content analysis. Br J Anaesth. 2012 Jul;109(1):99-109. doi: 10.1093/bja/aes184. PMID 22696559
- [Result] Lucisano KE, Talbot LA. Simulation training for advanced airway management for anesthesia and other healthcare providers: a systematic review. AANA J. 2012 Feb;80(1):25-31. PMID 22474801
- [Result] Chilkoti G, Mohta M, Wadhwa R, Saxena AK. Problem-based learning research in anesthesia teaching: current status and future perspective. Anesthesiol Res Pract. 2014;2014:263948. doi: 10.1155/2014/263948. Epub 2014 May 29. PMID 24982673
- [Result] Lui PW. Things we should know when designing simulator-based teaching in difficult airway management. J Chin Med Assoc. 2008 Apr;71(4):163-5. doi: 10.1016/S1726-4901(08)70098-4. No abstract available. PMID 18436497
- [Result] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266
- [Result] Langeron O, Cuvillon P, Ibanez-Esteve C, Lenfant F, Riou B, Le Manach Y. Prediction of difficult tracheal intubation: time for a paradigm change. Anesthesiology. 2012 Dec;117(6):1223-33. doi: 10.1097/ALN.0b013e31827537cb. PMID 23135259
- [Result] Cook TM, Woodall N, Harper J, Benger J; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 2: intensive care and emergency departments. Br J Anaesth. 2011 May;106(5):632-42. doi: 10.1093/bja/aer059. Epub 2011 Mar 29. PMID 21447489
- [Result] Vuori M, Akila R, Kalakoski V, Pentti J, Kivimaki M, Vahtera J, Harma M, Puttonen S. Association between exposure to work stressors and cognitive performance. J Occup Environ Med. 2014 Apr;56(4):354-60. doi: 10.1097/JOM.0000000000000129. PMID 24709760